CLINICAL TRIAL: NCT06117540
Title: An Open-label, Single-arm, Multicenter Phase II Clinical Study to Evaluate the Efficacy and Safety of WX390 in Patients With Advanced Solid Tumors
Brief Title: A Study of WX390 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WX390-002
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WX390 (Experimental): Participants will receive WX390 continuous oral dosing (1.1 mg once a day).
  Interventions: Drug: WX390

INTERVENTIONS:
Drug: WX390 — WX390 tablet, 1.1 mg once a day
  Other Names: WXFL10030390

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of WX390 in patients with advanced solid tumors. The main questions it aims to answer are:

* PFS, OS, DoR at week 48;
* antitumor effects at week 24 and week 48. Participants will be treated with WX390 orally, and follow the efficacy and safety evaluation according to the protocol.

DETAILED DESCRIPTION:
This study will be an open-label, multicenter phase II clinical trial. After being informed about the study and potential risks, all patients giving written informed consent will undergo a 4-week screening period to determine eligibility for study entry. And then patents will be administered for 12 cycles treatment and 30 days safety follow up after the last dose of treatment. The efficacy and safety measures will be conducted and collected every cycle.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Histological or cytological confirmed advanced solid tumor, standard regimen failed
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy of more than 3 months
* At least one measurable lesion according to RECIST 1.1
* Adequate organ function
* Signed and dated informed consent

Exclusion Criteria:

* Anti-cancer therapy within 30 days prior to the initiation of investigational treatment
* Major surgery within 30 days prior to the initiation of study treatment
* Toxicity from a previous anti-tumor treatment that does not return to Grade 0 or 1 (except for alopecia)
* Patients who are suffering active interstitial lung disease
* Evidence of ongoing or active serious infection
* Received corticosteroids treatment or other immunodepressant within 2 weeks before the first dose of study treatment
* Active hepatitis B or C infection
* Inability to take medication orally
* Abuse of alcohol or drugs
* Pregnant or lactating women
* People with cognitive and psychological abnormality or with low compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2025-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Week 48
  PFS, time from the first dose of trial medication to the first occurrence of disease progression or death due to any cause on study, whichever occurs first.
Overall Survival (OS) | Week 48
  OS, time from first dose of trial medication to death due to any cause.
Duration of Response (DOR) | Week 48
  DoR, the time from the first occurrence of objective response until disease progression or death from any cause, whichever occurs first.
Progression-free survival rate (PFSR) | Week 24 and Week 48
  PFSR, Percentage of patients alive without progression from baseline.
Objective Response Rate (ORR) | Week 24 and Week 48
  ORR, proportion of patients with complete response (CR) or partial response (PR).
Disease control rate (DCR) | Week 24 and Week 48
  DCR, proportion of patients with CR or PR or SD.

SECONDARY OUTCOMES:
Incidence, nature, and severity of adverse events (AEs) | Week 24 and Week 48
  Incidence, nature, and severity of adverse events (AEs) refer to the frequency, type, and level of harm of undesirable effects in clinical trials. Incidence shows how often AEs occur. Nature describes the specific characteristics of AEs, while severity indicates the extent of harm caused.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China